CLINICAL TRIAL: NCT05034965
Title: Dynamic Changes in Some Facial Muscles After Superficial Versus Deep Hyaluronic Acid Injection: An Electromyographic Study
Brief Title: Dynamic Changes in Some Facial Muscles After Hyaluronic Acid Filler Injection
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, marwa eldeeb, lecturer of dermatology, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0106665
Record Dates: First submitted 2021-08-28; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Changes in Facial Muscles Following Filler Injection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep injection of hyaluronic acid fillers (Active Comparator): Each female will receive filler injection deep to the muscle (supraperiosteal) on one side of the face.
  Interventions: Drug: hyaluronic acid filler injection
- superficial injection of hyaluronic acid fillers (Active Comparator): Each female will receive filler injection at superficial level to the muscle (subcutaneous) on the contralateral side(same dose and same site).
  Interventions: Drug: hyaluronic acid filler injection

INTERVENTIONS:
Drug: hyaluronic acid filler injection — quantitative surface electromyography before injection(baseline) and one week after injection
  Other Names: quantitative surface electromyography

SUMMARY:
assess electrophysiological changes in some facial muscle dynamics following hyaluronic acid filler injection in superficial versus deep level of injection.

DETAILED DESCRIPTION:
Participants will be subjected to injection of cross-linked hyaluronic acid fillers on both sides of the face in 3 different regions: temples, cheeks and chins.

Each female will undergo:

1. Before injection:

   1. Aesthetic facial clinical analysis.
   2. Baseline quantitative surface electromyography.
   3. Baseline digital photography.
2. Injection:

   Each female will receive the injection in the particular facial region at superficial level to the muscle (subcutaneous) on one side and the same amount at deep level to the muscle (supraperiosteal) on the other side.
3. One week after injection:

   1. Follow up quantitative surface electromyography.
   2. Follow up digital photography.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-60 years.
2. Sex: females.
3. Areas eligible for injection: temples, cheeks and chin.

Exclusion Criteria:

1. Active infection near the site of injection.
2. Pregnant or lactating women.
3. Patients suffering from any neuromuscular disorders.
4. Known allergy/hypersensitivity to hyaluronic acid fillers.
5. History of botulinum toxin injection in the last 4 months.
6. History of injection of fillers in the last 2 years.
7. Patients receiving any muscle relaxants.
8. Coagulation disorder or anticoagulants therapy.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
electrophysiological changes in some facial muscles | one week
  baseline and follow up quantitative surface electromyography

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt